CLINICAL TRIAL: NCT04237207
Title: Evaluation of AutoSense OS on a Cochlear Implant Sound Processor Programmed With Target CI Fitting Software in Adult Users of the HiResolution Bionic Ear System
Brief Title: Clinical Evaluation of a Cochlear Implant Sound Processor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR1218
Record Dates: First submitted 2020-01-07; First posted 2020-01-23 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-04

CONDITIONS: Hearing Loss; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases
MeSH Terms: conditions — Hearing Loss; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Aidable Residual Hearing (ARH) Cohort (Other): Control Device followed by experimental Device.
  Interventions: Device: Naída Cochlear Implant Q90 sound processor (Naida CI Q90) & software; Device: 301-M062 sound processor & software
- Electric Only (EO) Cohort (Other): Control Device followed by experimental Device.
  Interventions: Device: Naída Cochlear Implant Q90 sound processor (Naida CI Q90) & software; Device: 301-M062 sound processor & software

INTERVENTIONS:
Device: Naída Cochlear Implant Q90 sound processor (Naida CI Q90) & software — Control cochlear implant sound processor
Device: 301-M062 sound processor & software — New cochlear implant sound processor

SUMMARY:
This is a prospective within-subjects repeated-measures study that will enroll 24 adult users implanted with a HiResolution Bionic Ear System (HiRes 90K or newer). Subjects will be assigned to one of two cohorts based on audiometric results at the Baseline visit

DETAILED DESCRIPTION:
The overall goal of this clinical study is to demonstrate the safety and efficacy of a cochlear implant sound processor. Hearing outcomes are expected to be similar non-inferior to as compared to the currently approved software and processors. Therefore, the study described herein uses a non-inferiority design to determine whether sentence recognition in quiet and in noise is no worse with the new sound processor than with currently approved software on a Q90 processor.

ELIGIBILITY:
General Inclusion Criteria:

* Ability to provide Informed Consent
* 18 years of age or older
* Unilateral user of a HiResolutionTM Bionic Ear System (HiRes 90KTM, HiRes 90KTM Advantage, HiResTM Ultra, HiResTM Ultra 3D), including bilaterally implanted subjects that only use one implant in their everyday listening modality
* Minimum of 6 months of CI experience
* Having used a Naída CI Q70 or a Naída CI Q90 as their primary processor for a minimum of one month
* Presently using a current steering strategy
* At least moderate open-set speech recognition abilities with implant alone, as defined by achieving a score of ≥ 60% words correct in the AzBio in quiet test using the Naída CI Q90 research processor
* English language proficiency as determined by the investigator
* Willingness to use a BTE processor for the duration of the study

ARH Arm Inclusion Criteria

* Residual low frequency hearing sensitivity (pure tone average of < 70 dB HL for 125, 250, and 500 Hz) and a severe-to-profound high-frequency sensorineural hearing loss (pure tone average of ≥ 70 dB HL for 1,000, 2,000, 3000, 4,000, and 8,000 Hz) in the implanted ear
* Willingness to use an in-canal acoustic earhook for the duration of the study

EO Arm Inclusion Criteria

• Severe-to-profound sensorineural hearing loss in the low (pure tone average of ≥ 70 dB HL for 125, 250, and 500 Hz) and high frequencies (pure tone average ≥ 70 dB HL for 1,000, 2,000, 3000, 4,000, and 8,000 Hz) in the implanted ear

Exclusion Criteria:

* Unrealistic expectations regarding potential benefits, risks and limitations of the investigational device as determined by the investigator
* Unwillingness or physical / cognitive inability of subject to comply with all investigational requirements as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Tampa Bay Hearing and Balance Center, Tampa, Florida
  - Midwest Ear Institute/St. Luke's Health System, Kansas City, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Ear, Nose & Throat Clinic, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators recruited study subjects from their clinical practices. The first patient first visit occurred on December 17, 2019 and last patient last visit occurred on October 15, 2020. A total of 22 subjects were enrolled; 10 subjects were enrolled in the Electric Only cohort and 12 subjects were enrolled in the Aidable Residual Hearing cohort based on the results of their audiometric testing. All 22 subjects completed the study; there were no withdrawals or losses to follow-up.
Pre-assignment Details: After undergoing the Informed Consent Form process, subjects completed audiometric testing and speech perception testing to determine eligibility and assignment to either the electric only (EO) or aidable residual hearing (ARH) cohort. Subjects that did not meet the audiometric threshold hearing or speech testing inclusion criteria were discontinued at baseline.
Groups:
- Electric Only (EO) Cohort: Control Device followed by experimental Device.
  Naída Cochlear Implant Q90 (Naída CI Q90) sound processor & software: Control cochlear implant sound processor
  301-M062 sound processor & software: New cochlear implant sound processor
- Aidable Residual Hearing (ARH) Cohort: Control Device followed by experimental Device.
  Naída Cochlea Implant Q90 (Naída CI Q90) sound processor & software: Control cochlear implant sound processor
  301-M062 sound processor & software: New cochlear implant sound processor
Period: Overall Study
Arm/Group | Electric Only (EO) Cohort | Aidable Residual Hearing (ARH) Cohort
Started | 10 (Due to differences in speed of enrollment between the two cohorts and the delay in enrollment due to the Coronavirus (COVID-19) pandemic, enrollment for the electric only cohort was capped at 10 subjects, which exceeds the minimum sample size of 8 subjects per cohort.) | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subject assigned to ARH cohort were residual low frequency hearing sensitivity (PTA of < 70 dB HL for 125 thru 500 Hz) and a severe-to-profound high-frequency sensorineural hearing loss (pure tone average of ≥ 70 dB HL for 1000 thru 8000 Hz) in the implanted ear. EO cohort assigned to subjects with Severe-to-profound sensorineural hearing loss in the low (pure tone average of ≥ 70 dB HL for 125 thru 500 Hz) and high frequencies (PTA ≥ 70 dB HL for 1000 thru 8000 Hz) in the implanted ear
Groups:
- Aidable Residual Hearing (ARH) Cohort; Electric Only (EO) Cohort: Control Device followed by experimental Device.
  Naída Cochlear Implant Q90 (Naída CI Q90) sound processor & software: Control cochlear implant sound processor
  301-M062 sound processor & software: New cochlear implant sound processor
- Total: Total of all reporting groups
Arm/Group | Aidable Residual Hearing (ARH) Cohort | Electric Only (EO) Cohort | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants] — Population: Three subjects failed ARH baseline and 1 failed EO baseline.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 6 | 3 | 9
    >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Three subjects failed ARH baseline and 1 failed EO baseline.
  years | 61.1 (9.66) | 67.2 (9.28) | 64.5 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Three subjects failed ARH baseline and 1 failed EO baseline.
  Participants
    Female | 9 | 5 | 14
    Male | 3 | 5 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Three subjects failed ARH baseline and 1 failed EO baseline.
  participants
    United States | 12 | 10 | 22
Audiometric Threshold Testing and Speech Perception Testing [Count of Participants; unit: Participants] — A sample size of 12 subjects per cohort was calculated based upon the primary efficacy outcomes measure i.e., demonstration of non-inferiority of AutoSense on the M90 process compared to AutoSound on the Q90 processor. The calculations were based on 8 complete subjects per cohort, with a total of 12 subjects enrolled in order to accommodate up to 4 subjects per cohort who may have screen failed or early discontinued. Population: Four subjects did not meet inclusion criteria and were therefore discontinued at baseline.
  Participants | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Speech Recognition in Quiet
Description: The primary efficacy endpoints are AzBio sentence recognition scores in quiet at Baseline with the new sound processor as compared to AzBio sentence recognition scores in quiet at Baseline with currently approved software on a Q90 processor. Scores are determined on a scale of 0% to 100% words correct with higher scores indicating a better outcome.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: percentage of correct words
Groups:
- EO Cohort; ARH Cohort: Control Device followed by experimental Device.
  Naída CI Q90 sound processor & software: Control cochlear implant sound processor
  301-M062 sound processor & software: New cochlear implant sound processor
Arm/Group | EO Cohort | ARH Cohort
Number analyzed (Participants) | 10 | 12
percentage of correct words
  Baseline AutoSound | 88.31 (5.817) | 89.39 (10.535)
  Baseline AutoSense | 87.30 (10.214) | 88.09 (9.848)
Statistical Analysis 1: Comparison: EO Cohort vs ARH Cohort; Test type: Non-Inferiority — The primary efficacy objective is to demonstrate non-inferiority of AutoSense on the M90 processor compared to AutoSound on the Q90 processor for the AzBio sentence test in quiet mode based on a paired t-test. The primary efficacy analyses will test the null hypothesis (inferiority) that the mean of the paired differences in AzBio sentence scores in quiet mode (AutoSense on M90 - AutoSound on Q90) are less than or equal to -10 percentage points; p = 0.0010, t-test, 2 sided

2. Secondary Outcome: Speech Recognition in Noise
Description: Demonstrate that AzBio sentence recognition scores in noise with the new sound processor are no worse than AzBio sentence recognition scores in noise with currently approved software on a Q90 processor. Scores are determined on a scale of 0% to 100% words correct with higher scores indicating a better outcome.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: percentage of correct word responses
Arm/Group | EO Cohort | ARH Cohort
Number analyzed (Participants) | 10 | 12
percentage of correct word responses
  AutoSound | 52.95 (31.163) | 66.04 (25.939)
  AutoSense | 76.37 (19.078) | 84.98 (13.108)
Statistical Analysis 1: Comparison: EO Cohort vs ARH Cohort; Test type: Non-Inferiority — The 1st secondary endpoint was to demonstrate that speech recognition in noise with AutoSense on a 301-M062 processor was no worse than speech recognition in noise with currently approved software on a Q90 processor; p = 0.0010, t-test, 2 sided

3. Secondary Outcome: Increased Speech Recognition in Noise
Description: Demonstrate increased AzBio sentence recognition scores in noise with the new sound processor when comparing "Omnidirectional" program to AutoSense. Omnidirectional refers to a setting in which the AutoSense feature is not active. Scores are determined on a scale of 0% to 100% words correct with higher scores indicating a better outcome.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: percentage of correct words recognized
Arm/Group | EO Cohort | ARH Cohort
Number analyzed (Participants) | 10 | 12
percentage of correct words recognized
  Omnidirectional | 42.93 (30.801) | 51.37 (28.604)
  AutoSense | 76.37 (19.078) | 84.98 (13.108)
Statistical Analysis 1: Comparison: EO Cohort vs ARH Cohort; Test type: Non-Inferiority — The 2nd secondary endpoint was to demonstrate increased speech recognition in noise with the 301-M062 sound processor when comparing "Omnidirectional" program to AutoSense; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: AEs were recorded and tracked between completion of the informed consent form (signed and dated) and two weeks after the participant's last study visit. The total period is up to 5 weeks.
Description: All device-related and non-device-related adverse events (AEs) was tracked and reported accordingly throughout the study as defined in the investigational plan and in accordance with requirements of an IDE investigation. The number and percent of all subjects experiencing adverse events was summarized by type, status and frequency of event.
Arm/Group | EO Cohort | ARH Cohort
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 2/10 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EO Cohort (N=10) | ARH Cohort (N=12)
Patient discomfort (Product Issues) | 0 (0) | 1 (1) — Participant reported sharpness of sound that was sometimes uncomfortable and sound was distorted.
Upper Respiratory (Infections and infestations) | 1 (1) | 0 (0) — Subject reported a head cold
Sprained ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject twisted ankle playing golf.

LIMITATIONS AND CAVEATS:
Due to clinic closures related to the COVID-19 pandemic, total enrollment in the EO Cohort was 10 subjects instead of 12.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees to submit any publication to Sponsor at least 30 days before submission. Within 30 days of its receipt, Sponsor advises PI in writing of any information contained therein which is Confidential Information (other than Study Data) or which may impair availability of patent protection for Inventions. Sponsor has the right to require PI to remove specifically identified CI and/or to delay the publication for an additional 60 days to enable Sponsor to seek patent protection for Inventions.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT04237207/Prot_SAP_000.pdf